CLINICAL TRIAL: NCT04579094
Title: Prevalence and Risk Factors for the Carriage of Multi- and Highly Resistant Bacteria and Clostridioid Difficile Toxigenic in Residents and Healthcare Workers in Nursing Home (PREMS)
Brief Title: Prevalence and Risk Factors for the Carriage of Bacteria and Clostridioid in Elderly Dependent Persons
Acronym: PREMS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2019/JO-01
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Elderly; Healthcare Associated Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/elderly dependent persons
  Interventions: Other: Feces sampling at inclusion (J0)
- 2/healthcare workers (HCW)
  Interventions: Other: Feces sampling at inclusion (J0)

INTERVENTIONS:
Other: Feces sampling at inclusion (J0) — Feces sampling at inclusion (J0)

SUMMARY:
Brief summary : Very few studies have evaluated the prevalence of multi-drug resistant (MDR), highly resistant emerging bacteria and Clostridioides difficile toxinogenic (CDt) in residents and in healthcare workers (HCW) in nursing home (NH). Most of study were conducted in acute care services and were limited to specific bacterial species.

Hypothesis : The carriage of MDR bacteria in resident may be a risk factor for an outbreak in NH or in healthcare facility.

Primary outcome: The objective of this study is to estimate the prevalence for carriage of MDR bacteria and CDt in residents in NH.

Secondary outcomes:

* Estimate the prevalence for carriage of MDR bacteria and CDt toxigenic in HCW in NH.
* Identify the risk factors for carriage of MDR bacteria and CDt in residents in nursing home
* Identify the risk factors for carriage of MDR bacteria and CDt in healthcare workers in NH
* Evaluate the presence of cross-transmission of MDR bacteria and CDt in one or several NH
* Evaluate the association between the presence of cross-transmission of MDR bacteria and CDt in a NH and the management of infection control
* Establishment a collection of stool samples

ELIGIBILITY:
* Inclusion criteria:
* Resident :

The resident must be a member or beneficiary of a health insurance. The resident is in permanent accommodation whose the date of admission is at least 1 month earlier on the day of collection.

* healthcare workers : The healthcare workers must be a member or beneficiary of a health insurance. The healthcare workers begin to work in nursing at least 1 month earlier on the day of collection.
* Exclusion criteria:
* Resident :

The resident refuses to participate.

o healthcare workers : The healthcare workers refuses to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of the study is all elderly residents of nursing home and their caregivers. The source population of the study corresponds to the residents of the 61 nursing home in the Gard region, and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Presence or absence of multi-drug resistant bacteria in residents' feces. | at inclusion (J0)
  prevalence of carriage of multi-drug resistant bacteria
Presence or absence of Highly Resistant and Emerging Bacteria in residents' feces. | at inclusion (J0)
  prevalence of carriage of Highly Resistant and Emerging Bacteria
Presence or absence of Clostridioids difficult toxinogenic in residents' feces. | at inclusion (J0)
  prevalence of carriage of Clostridioids difficult toxinogenic

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Hôpital Universitaire Carémeau, Nîmes, France